CLINICAL TRIAL: NCT04577066
Title: Safety and Protective Efficacy of Genetically Attenuated Pf∆mei2 (Also Referred to as GA2) Malaria Parasites in Healthy Dutch Volunteers.
Brief Title: Safety and Preliminary Protective Efficacy of Genetically Attenuated GA2 Parasites.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Meta Roestenberg, Principal Investigator, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GA2
Record Dates: First submitted 2020-09-22; First posted 2020-10-06 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Plasmodium Falciparum Malaria
Keywords: Malaria; Plasmodium falciparum; Genetically attenuated parasites
MeSH Terms: conditions — Malaria, Falciparum; Malaria

STUDY DESIGN:
Intervention Model Description: This trial has both a sequential as well as a parallel interventional study model.
  The safety and tolerability of the GA2 parasite will be assessed in phase 1 by means of a sequential study model. There will be 2 cohorts, which will be recruited sequentially and exposed to increasing numbers of infected mosquito bites.
  The preliminary protective efficacy of the GA2 parasite will be assessed in phase 2 by means of a parallel study model. There will be 3 groups of volunteers, who will be exposed to either GA2-infected, GA1-infected or uninfected mosquito bites.
Who Masked: Participant, Investigator
Masking Description: Phase 1 will be an open label trial, Phase 2 will be a double-blind trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (GA2) (Experimental): Volunteers will be exposed to GA2-infected mosquito bites.
  Interventions: Other: GA2
- Group 2 (GA1) (Active Comparator): Volunteers will be exposed to the GA1-infected mosquito bites.
  Interventions: Other: GA1
- Group 3 (Placebo) (Placebo Comparator): Volunteers will be exposed to uninfected mosquito bites.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: GA2 — 15 volunteers will receive 50 GA2-infected mosquito bites. The GA2 parasite is a new genetically attenuated Plasmodium falciparum parasite, which arrests development in the liver and should not be able to cause malaria in humans.
  Arms: Group 1 (GA2)
Other: GA1 — 10 volunteers will receive 50 GA1-infected mosquito bites. The GA1 parasite is a genetically attenuated Plasmodium falciparum parasite, which arrests development in the liver and is not able to cause malaria in humans.
  Arms: Group 2 (GA1)
Other: Placebo — 5 volunteers will receive 50 uninfected mosquito bites.
  Arms: Group 3 (Placebo)

SUMMARY:
This study will consist of two phases and be aimed at assessing the safety and tolerability of the new genetically attenuated GA2 malaria parasite (Phase 1) and its preliminary protective efficacy against controlled human malaria infection (Phase 2) in healthy Dutch volunteers.

DETAILED DESCRIPTION:
Malaria is one of the most common tropical diseases, accounting for 228 million infections and 450.000 deaths each year. It is caused by five species of protozoan parasites belonging to the genus of the Plasmodia. Plasmodia have a complex life cycle: they are injected into the human host by female Anopheles mosquitos, migrate to the liver to replicate and then enter red blood cells. The typical symptoms of malaria with fever episodes are caused by the bursting of red blood cells, as the parasites leave to infect new cells.

The rising resistance of both parasites against anti-malarial drugs and mosquitoes against insecticides, make the need to eradicate malaria even more impellent. A promising approach to disease control is the development of an effective vaccine. Among the different approaches to vaccine development, live attenuated parasites stand out for their high protective efficacy (>90%).

The GA2 parasite, a new genetically attenuated malaria parasite, which is derived from the NF45 Plasmodium falciparum strain and has been engineered to arrest development in the liver before entering the bloodstream, was recently created. It should therefore not be able to cause malaria in humans. The idea is that the GA2 parasite will prime the immune system for recognition of non attenuated parasites in the future without causing disease itself. In other words, exposure to the innocuous GA2 parasite could confer protection against pathogenic malaria parasites.

Hence, this study is aimed at investigating the safety and tolerability of the GA2 parasite and at determining its potential protective efficacy against controlled human malaria infection. The former question will be investigated by exposing volunteers to sequentially increasing numbers of GA2-infected mosquito bites. The latter question will be investigated by repeatedly (3 times) exposing volunteers to the GA2 parasite and once to unattenuated parasites. The efficacy of the GA2 parasite will be compared to another genetically attenuated parasite, the GA1, which in previous studies has been shown to be safe and well-tolerated but only have limited protective efficacy. There will also be a placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Subject is aged ≥ 18 and ≤ 35 years and in good health.
* Subject has adequate understanding of the procedures of the study and agrees to abide strictly thereby.
* Subject is able to communicate well with the investigator, is available to attend all study visits.
* Furthermore, the subject will remain within the Netherlands from day -1 till day +28 after each parasite exposure. After CHMI, subjects have to be reachable by phone (24/7) from day -1 until day 35.
* Subject agrees to inform his/her general practitioner (GP) about participation in the study.
* Subject agrees to refrain from blood donation to Sanquin or for other purposes throughout the study period and for a defined period thereafter according to Sanquin guidelines.
* Non-pregnant, non-lactating females of reproductive potential (i.e., have a uterus and are neither surgically sterilized nor post-menopausal) agree to use adequate contraception and to not breastfeed for the duration of study.
* Subject agrees to refrain from intensive physical exercise (disproportionate to the subjects' usual daily activity or exercise routine) for twenty-one days following each immunization and during the malaria challenge period.

Exclusion Criteria:

* Any history, or evidence at screening, of clinically significant symptoms, physical signs or abnormal laboratory values suggestive of systemic conditions, such as cardiovascular, pulmonary, renal, hepatic, neurological, dermatological, endocrine, malignant, hematological, infectious, immune-deficient, psychiatric or other disorders, which could compromise the health of the volunteer during the study or interfere with the interpretation of the study results. These include, but are not limited to, any of the following:

  a. Body weight <50 kg or Body Mass Index (BMI) <18.0 or >30.0 kg/m2 at screening.

  b. A heightened risk of cardiovascular disease, defined as: An estimated ten-year risk of fatal cardiovascular disease of ≥5% at screening, as determined by the Systematic Coronary Risk Evaluation (SCORE); i. An estimated ten-year risk of fatal cardiovascular disease of ≥5% at screening, as determined by the Systematic Coronary Risk Evaluation (SCORE); ii. History, or evidence at screening, of clinically significant arrhythmia's, prolonged QT-interval or other clinically relevant ECG abnormalities; or iii. A positive family history of cardiac events in first or second degree relatives (according to the system used in medical genetics) <50 years old.

  c. Functional asplenia, sickle cell trait/disease, thalassemia trait/disease or G6PD deficiency.

  d. History of epilepsy in the period of five years prior to study onset, even if no longer on medication.

  e. Positive HIV, HBV or HCV screening tests. f. Chronic use of i) immunosuppressive drugs, ii) antibiotics, iii) or other drugs that might have an influence on the immune system (excluding inhaled and topical corticosteroids and incidental use of oral anti-histamines), within three months prior to study onset or expected use of such during the study period.

  g. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past five years.

  h. Any history of treatment for severe psychiatric disease by a psychiatrist in the past year.

  i. History of drug or alcohol abuse interfering with normal social function in the period of one year prior to study onset, positive urine toxicology test for cocaine, amphetamines or cannabis at screening.
* For female subjects: breastfeeding, or positive urine pregnancy test at screening or prior to immunization or prior to CHMI.
* Any history of malaria, positive serology for Pf, or previous participation in any malaria (vaccine) study or CHMI.
* Known hypersensitivity to or contra-indications (including co-medication) for use of atovaquone/proguanil or artemether/lumefantrine, or history of severe (allergic) reactions to MB.
* Receipt of any vaccinations in the three months prior to the start of the study or plans to receive any other vaccinations during the study period or up to eight weeks thereafter. Exceptions are made for influenza vaccination and for vaccination against the coronavirus SARS-COV2 or any other vaccination which cannot be reasonably withheld or postponed.
* Participation in any other clinical study in the 30 days prior to the start of the study or during the study period.
* Being an employee or student of the department of Parasitology, Medical Microbiology or Infectious Diseases of the RadboudUMC or the LUMC.
* Any other condition or situation that would, in the opinion of the investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol or would compromise the integrity of the data.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Number of volunteers with blood-stage parasitemia. | From time of exposure to 28 days later.
  The number of volunteers developing a breakthrough blood-stage infection after exposure to the GA2 parasite will be calculated as absolute numbers. Frequencies will be calculated by dividing the number of qPCR positive volunteers by the total number of volunteers in each group and multiplying the result by 100.
Number of volunteers protected against controlled human malaria infection immunisation with the GA2 parasite. | From first immunisation to 104 days later.
  The number of volunteers protected against CHMI in each group will be calculated as absolute numbers. Frequencies will be calculated by dividing the number of qPCR positive volunteers by the total number of volunteers in each group and multiplying the result by 100. The difference between the intervention group (receiving bites of GA2-infected mosquitoes) and control group (receiving bites of uninfected mosquitoes) will be calculated by means of the Chi square test.
Number and magnitude of adverse events in Phase 1 and Phase 2. | From exposure to maximum 264 days later.
  The number of graded adverse events occurring in each group will be calculated as absolute numbers. Frequencies will be calculated by dividing the number of graded adverse events occurring in each group by the total number of volunteers in each group.

SECONDARY OUTCOMES:
Humoral immune responses of volunteers exposed to the GA2 and GA1 parasite. | From time of exposure to maximum 264 days later.
  Difference in concentration of anti-CSP antibodies between GA2 and GA1 immunised volunteers as assessed by ELISA prior to controlled human infection (study day 75).
Cellular immune response of volunteers exposed to the GA2 and GA1 parasite. | From time of exposure to maximum 264 days later.
  Difference in percentage of CD4+ and CD8+ T-cells producing IFN-γ between GA2 and GA1 immunised volunteers as assessed by flow cytometry prior tot controlled human infection (study day 75).

CONTACTS AND LOCATIONS:
Overall Officials: Meta Roestenberg, MD, PhD, Prof., Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

REFERENCES:
- [Background] Ashley EA, Pyae Phyo A, Woodrow CJ. Malaria. Lancet. 2018 Apr 21;391(10130):1608-1621. doi: 10.1016/S0140-6736(18)30324-6. Epub 2018 Apr 6. PMID 29631781
- [Background] Hoffman SL, Goh LM, Luke TC, Schneider I, Le TP, Doolan DL, Sacci J, de la Vega P, Dowler M, Paul C, Gordon DM, Stoute JA, Church LW, Sedegah M, Heppner DG, Ballou WR, Richie TL. Protection of humans against malaria by immunization with radiation-attenuated Plasmodium falciparum sporozoites. J Infect Dis. 2002 Apr 15;185(8):1155-64. doi: 10.1086/339409. Epub 2002 Apr 1. PMID 11930326
- [Background] Roestenberg M, McCall M, Hopman J, Wiersma J, Luty AJ, van Gemert GJ, van de Vegte-Bolmer M, van Schaijk B, Teelen K, Arens T, Spaarman L, de Mast Q, Roeffen W, Snounou G, Renia L, van der Ven A, Hermsen CC, Sauerwein R. Protection against a malaria challenge by sporozoite inoculation. N Engl J Med. 2009 Jul 30;361(5):468-77. doi: 10.1056/NEJMoa0805832. PMID 19641203
- [Derived] Lamers OAC, Franke-Fayard BMD, Koopman JPR, Roozen GVT, Janse JJ, Chevalley-Maurel SC, Geurten FJA, de Bes-Roeleveld HM, Iliopoulou E, Colstrup E, Wessels E, van Gemert GJ, van de Vegte-Bolmer M, Graumans W, Stoter TR, Mordmuller BG, Houlder EL, Bousema T, Murugan R, McCall MBB, Janse CJ, Roestenberg M. Safety and Efficacy of Immunization with a Late-Liver-Stage Attenuated Malaria Parasite. N Engl J Med. 2024 Nov 21;391(20):1913-1923. doi: 10.1056/NEJMoa2313892. PMID 39565990